CLINICAL TRIAL: NCT05963152
Title: The Effects of Resistance Exercise on Cognition in People With Type 1 Diabetes: a Randomised Controlled Trial
Brief Title: Resistance Exercise and Cognition in People With Type 1 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dasman Diabetes Institute (Other)
Responsible Party: Principal Investigator, Dr. Ebaa Al Ozairi, Chief Medical Officer, Dasman Diabetes Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RA HM-2023-010
Record Dates: First submitted 2023-07-07; First posted 2023-07-27 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: type1diabetes
Keywords: exercise; cognition
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: 1:1:1 parallel group design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): Habitual Physical Activity
  Interventions: Behavioral: Habitual Physical Activity
- Morning exercise (Experimental): Exercise training between 6-10am
  Interventions: Behavioral: Morning Exercise
- Afternoon exercise (Experimental): Exercise training between 4-8pm
  Interventions: Behavioral: Afternoon Exercise

INTERVENTIONS:
Behavioral: Habitual Physical Activity — Participants will be asked to maintain their normal activity levels
  Arms: Control
Behavioral: Morning Exercise — Between 6-10am participants will attend the gym and perform 10 min of warm up exercise, 3 sets of 7 resistance exercises ( leg press, calf press, leg curl, chest press, lateral raise, seated row and plank)
  Arms: Morning exercise
Behavioral: Afternoon Exercise — Between 4-8pm participants will attend the gym and perform 10 min of warm up exercise, 3 sets of 7 resistance exercises ( leg press, calf press, leg curl, chest press, lateral raise, seated row and plank)
  Arms: Afternoon exercise

SUMMARY:
The aim of the current study is to determine the effects of resistance exercise on performance of the Paced Auditory Serial Addition Test and the Colour Trails Test.

ELIGIBILITY:
Inclusion Criteria:

* Physician confirmed type 1 diabetes for at least 1 year
* Stable insulin therapy for 3 months prior to the study

Exclusion Criteria:

* BMI of 45 or higher
* BP of 160/100mmHg or higher
* autonomic neuropathy
* severe proliferative retinopathy
* joint or limb injuries preventing weight-bearing activity
* autonomic neuropathy
* severe proliferative retinopathy
* any other medical condition that prevents participants from exercising safely.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Chronic change in Paced Auditory Serial Addition Test (PASAT) score | Change from baseline to 12 weeks
  Measured using the standardised Paced Auditory Serial Addition Test (PASAT) score ranging from 0-60 with a higher score meaning a better outcome
Chronic change in Colour Trails Test score | Change from baseline to 12 weeks
  Measured using the standardised Colour Trails Test, with score based on completion time (0-240s), number of errors, error type, and number of prompts with a shorter completion time and lower number of errors and prompts indicating a better outcome

SECONDARY OUTCOMES:
Baseline acute change in Paced Auditory Serial Addition Test (PASAT) score | Change from before (0 hour) to 1 hour post exercise during week 1
  Measured using the standardised Paced Auditory Serial Addition Test (PASAT) during the first exercise session, score ranging from 0-60 with a higher score meaning a better outcome
12 week acute change in Paced Auditory Serial Addition Test (PASAT) score | Change from before (0 hour) to 1 hour post exercise during week 12
  Measured using the standardised Paced Auditory Serial Addition Test (PASAT) during the last exercise session, score ranging from 0-60 with a higher score meaning a better outcome
Baseline acute change in Colour Trails Test score | Change from before (0 hour) to 1 hour post exercise during week 1
  Measured using the standardised Colour Trails Test during the first exercise session, with score based on completion time (0-240s), number of errors, error type, and number of prompts with a shorter completion time and lower number of errors and prompts indicating a better outcome
12 week acute change in Colour Trails Test score | Change from before (0 hour) to 1 hour post exercise during week 12
  Measured using the standardised Colour Trails Test during the last exercise session, with score based on completion time (0-240s), number of errors, error type, and number of prompts with a shorter completion time and lower number of errors and prompts indicating a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Dasman Diabetes Institute, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: No